CLINICAL TRIAL: NCT06830668
Title: Effectiveness and Persistence of Same-day Re-start with B/F/TAF Among Patients with HIV Who Experienced Discontinuation from Previous NNRTI Based Regimens in China
Brief Title: Same-Day Restart of B/F/TAF in HIV Patients After NNRTI Discontinuation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Center for AIDS/STD Control and Prevention, China CDC (Other Government)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-US-380-7381
Record Dates: First submitted 2025-01-26; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: HIV Infection; HIV
Keywords: HIV; HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AIDS patients who discontinued NNRTI for more than 90 days (Experimental): HIV patients of any gender, older than 18 years of age, who have been off their prior NNRTI regimen for more than 90 days and who have an HIV-1 viral load greater than 50 copies/uL.In this study, eligible patients will restart treatment on the same day and receive B/F/TAF for one year.We will conduct follow-ups on the patients and carry out routine clinical tests.
  Interventions: Drug: Regimen：BIC+FTC+TAF

INTERVENTIONS:
Drug: Regimen：BIC+FTC+TAF — Same-day restart of "BIC+FTC+TAF" among HIV patients who experienced discontinuation from previous NNRTI-based regimens

SUMMARY:
In China, free first-line ART regimens typically consist of two nucleoside reverse transcriptase inhibitors (NRTIs) and a non-nucleoside reverse transcriptase inhibitor (NNRTI). As of the end of 2022, approximately 1.135 million individuals were receiving ART, achieving a coverage rate of 92.8%, largely due to participation in free treatment programs. However, around 36,000 patients have discontinued treatment, primarily due to side effects associated with Efavirenz (EFV), a common NNRTI. The challenges posed by side effects and resistance profiles of existing NNRTIs highlight the need for effective re-initiation of ART to improve overall treatment coverage. INSTIs, particularly B/F/TAF (Bictegravir/emtricitabine/tenofovir alafenamide), demonstrates effective viral suppression and a higher barrier to resistance than NNRTIs. B/F/TAF has shown efficacy in patients with resistance mutations, making it a strong candidate for same-day ART re-initiation, especially in resource-limited areas where genotypic resistance testing may be unavailable. This study aims to evaluate the feasibility and effectiveness of rapidly restarting B/F/TAF in patients with treatment interruptions from previous NNRTI regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18 years old or above.
* Discontinuation of previous NNRTI based regimen for more than 90 days.
* No known CrCl< 30mL/min or severe hepatic impairment.
* No known or suspected resistance to BIC.
* No known pregnancy

Exclusion Criteria:

••Patients who are pregnant.

* Patients who have abnormal liver and kidney function indicators(Child-pugh class C, CrCl< 30).Hepatitis virus co-infection does not serve as an exclusion criterion.
* Patients who have historic resistance test indicating drug resistant to BIC or baseline resistance test indicating resistance to BIC.
* Patients who are psychiatric illness or active tuberculosis co-infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy of re-initiation of B/F/TAF | From enrollment to the end of treatment at 24 weeks
  Evaluate the efficacy following the re-initiation of B/F/TAF as determined by the achievement of HIV-RNA undetectable (< 50 copies/ml).

SECONDARY OUTCOMES:
Drug resistance status | From enrollment to the end of treatment at 48 weeks
  Describe drug resistance status
The reasons for discontinuation of prior therapy | From enrollment to the end of treatment at 1 week
  Describe the reasons for discontinuation of prior therapy
The efficacy of B/F/TAF | From enrollment to the end of treatment at Week 12, Week24 and Week 48
  Evaluate the efficacy of B/F/TAF (achievement of HIV-1 RNA< 50 copies/ml and HIV-1 RNA < 200 copies/ml) among those participants rapidly restarting B/F/TAF
The persistence on B/F/TAF . | From enrollment to the end of treatment at 48 weeks
  Evaluate the persistence on B/F/TAF during the study period and describe the reasons for discontinuation of B/F/TAF if it happens.
The changes in parameters of quality of life and treatment satisfaction | From enrollment to the end of treatment at Week24 and Week 48
  Describe changes in parameters of quality of life and treatment satisfaction
The safety and tolerability on B/F/TAF | From enrollment to the end of treatment at 48 weeks
  Evaluate the safety and tolerability on B/F/TAF during the study period.
The emergence of drug resistance | From enrollment to the end of treatment at 48 weeks
  Describe the emergence of drug resistance developed during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for AlDS/STD Control and Prevention,China CDC,NO.155, Changbai Road,Changping District,Beijing, Chian, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No